CLINICAL TRIAL: NCT00611403
Title: Safety and Efficacy Study of Cyclosporine Ophthalmic Emulsion in Post-LASIK Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 192371-014
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Results first posted 2011-12-20 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-11

CONDITIONS: Dry Eye Syndromes
Keywords: LASIK
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- RESTASIS® (Active Comparator): Cyclosporine Ophthalmic Emulsion 0.05% (RESTASIS®)
  Interventions: Drug: Cyclosporine Ophthalmic Emulsion 0.05% (RESTASIS®)
- REFRESH ENDURA® (Active Comparator): Artificial Tears (REFRESH ENDURA®)
  Interventions: Drug: Artificial Tears REFRESH ENDURA®

INTERVENTIONS:
Drug: Cyclosporine Ophthalmic Emulsion 0.05% (RESTASIS®) — Cyclosporine Ophthalmic Emulsion 0.05% administered twice daily in each eye for 6 months following LASIK surgery
  Arms: RESTASIS®
Drug: Artificial Tears REFRESH ENDURA® — REFRESH ENDURA® administered twice daily in each eye for 6 months following LASIK surgery
  Arms: REFRESH ENDURA®

SUMMARY:
This study will evaluate the safety and efficacy of cyclosporine ophthalmic emulsion administered twice daily following LASIK surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for bilateral LASIK surgery
* Patient is in good general health
* Eye glasses prescription of -1 to -8

Exclusion Criteria:

* Significant Dry Eye
* Presence of eye disease
* Uncontrolled systemic disease

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2007-12; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase
Arm/Group | RESTASIS® | REFRESH ENDURA®
Started | 68 | 69
Completed | 62 | 58
Not Completed | 6 | 11
Period: Post Treatment Extension Phase
Arm/Group | RESTASIS® | REFRESH ENDURA®
Started | 26 (26 of 68 pts who received RESTASIS® in the Treatment Phase entered the Post Treatment Ext. Phase) | 25 (25 of 69 pts who received ENDURA® in the Treatment Phase entered the Post Treatment Extension Phase)
Completed | 22 | 24
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RESTASIS® | REFRESH ENDURA® | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Customized [Number; unit: participants]
  < 30 years | 19 | 21 | 40
  Between 30 and 40 years | 25 | 24 | 49
  > 40 years | 24 | 24 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 79
  Male | 25 | 33 | 58

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clinical Success at Month 6
Description: Percentage of patients with clinical success at month 6. Clinical success is defined as the percentage of patients with corneal sensitivity (the capability of the cornea to respond to stimulation) >= 50 millimeters in all regions of the study eye at month 6 of the Treatment Phase.
Time Frame: Month 6
Population: Modified Intent-to-Treat (mITT). The mITT population included all randomized and treated patients with a study eye having a corneal sensitivity measurement of < 25 mm in the 3 central regions of the eye on Day 2.
Measure: Number; unit: Percentage of Patients
Arm/Group | RESTASIS® | REFRESH ENDURA®
Number analyzed (Participants) | 42 | 43
Percentage of Patients | 64.3 | 58.1

2. Secondary Outcome: Change From Baseline in Keratocyte Density in the Anterior Flap of the Eyes at Month 6
Description: Change from baseline in keratocyte (specialized cells in the cornea activated after injury or inflammation) density (thickness) in the anterior flap of the eyes (better eye and worse eye) at month 6 of the Treatment Phase. A positive number change from baseline represents an increase in density (improvement). A negative number change from baseline represents a decrease in density (worsening).
Time Frame: Baseline, Month 6
Population: Intent-to-Treat (ITT). The ITT population includes all patients who started the study (randomized).
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter (cells/mm^3)
Arm/Group | RESTASIS® | REFRESH ENDURA®
Number analyzed (Participants) | 68 | 69
Cells per cubic millimeter (cells/mm^3)
  Better Eye: Baseline | 28095.7 (5303.28) | 26069.5 (4648.48)
  Better Eye: Change from Baseline at Month 6 | 901.6 (6117.69) | 1346.6 (5550.24)
  Worse Eye: Baseline | 26489.9 (5161.53) | 27480.6 (4854.00)
  Worse Eye: Change from Baseline at Month 6 | 3011.7 (7931.29) | -218.4 (5799.30)

3. Secondary Outcome: Change From Baseline in Goblet Cell Density of the Eyes at Month 6
Description: Change from baseline in goblet cell density of the eyes (better eye and worse eye) at month 6 of the Treatment Phase. Goblet cells are special cells in the eye that support a healthy tear film. A positive number change from baseline represents an increase in goblet cells (improvement).
Time Frame: Baseline, Month 6
Population: Intent-to-Treat (ITT). The ITT population includes all patients who started the study (randomized).
Measure: Median (Full Range); unit: Cells per square millimeter (cells/mm^2)
Arm/Group | RESTASIS® | REFRESH ENDURA®
Number analyzed (Participants) | 68 | 69
Cells per square millimeter (cells/mm^2)
  Better Eye: Baseline | 60.9 [0 to 291] | 59.7 [0 to 193]
  Better Eye: Change from Baseline at Month 6 | 30.9 [-284 to 115] | -3.1 [-145 to 222]
  Worse Eye: Baseline | 68.4 [0 to 276] | 79.2 [2 to 237]
  Worse Eye: Change from Baseline at Month 6 | 15.4 [-96 to 222] | 9.9 [-175 to 208]

ADVERSE EVENTS:
Arm/Group | RESTASIS® | REFRESH ENDURA®
Serious Adverse Events (participants affected / at risk) | 1/68 | 1/69
Other Adverse Events (participants affected / at risk) | 16/68 | 8/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RESTASIS® (N=68) | REFRESH ENDURA® (N=69)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Infected bites (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RESTASIS® (N=68) | REFRESH ENDURA® (N=69)
Seasonal allergy (Immune system disorders) | 10 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo